CLINICAL TRIAL: NCT02390219
Title: A Phase 3b, Open-Label Study to Evaluate Lumacaftor and Ivacaftor Combination Therapy in Subjects 12 Years and Older With Cystic Fibrosis and Advanced Lung Disease, Homozygous for the F508del-CFTR Mutation
Brief Title: Study to Evaluate Lumacaftor and Ivacaftor Combination Therapy in Subjects 12 Years and Older With Advanced Lung Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX14-809-106
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Results first posted 2017-11-01 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-10

CONDITIONS: Cystic Fibrosis; Advanced Lung Disease
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor; ivacaftor

ARMS (1):
- Lumacaftor/Ivacaftor combination (Experimental): Lumacaftor 400 milligram (mg) and ivacaftor 250 mg combination tablet orally twice daily for 24 weeks.
  Interventions: Drug: Lumacaftor; Drug: Ivacaftor

INTERVENTIONS:
Drug: Lumacaftor
  Other Names: VX-809
Drug: Ivacaftor
  Other Names: VX-770

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of LUM/IVA combination therapy in subjects 12 years and older with CF and advanced lung disease and who are homozygous for the F508del CFTR mutation

ELIGIBILITY:
Inclusion Criteria:

* Homozygous for the F508del-CFTR mutation; historical genotype must be documented in the participant's source documents.
* Percent predicted FEV1 <40 of adjusted for age, sex, and height at Screening

Exclusion Criteria:

* Participant currently receiving invasive mechanical ventilation.
* History of any comorbidity that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant
* Any clinically significant laboratory abnormalities at screening that would interfere with the study assessments or pose an undue risk for the subject
* A 12-lead electrocardiograms (ECG) demonstrating QTcF >450 msec at Screening
* History of solid organ or hematological transplantation
* History of alcohol or drug abuse in the past year
* Ongoing or prior participation in an investigational drug study (including studies investigating lumacaftor and/or ivacaftor) within 30 days of screening.
* Use of strong inhibitors, moderate inducers, or strong inducers of CYP3A
* Pregnant and nursing females: Females of childbearing potential must have a negative pregnancy test at Screening and Day 1.
* Sexually active subjects of reproductive potential who are not willing to follow the contraception requirements
* Use of beta blockers or the equivalent at Screening.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Denver, Colorado
  - Tampa, Florida
  - Chicago, Illinois
  - St Louis, Missouri
  - Pittsburgh, Pennsylvania
  - Houston, Texas

REFERENCES:
- [Derived] Taylor-Cousar JL, Jain M, Barto TL, Haddad T, Atkinson J, Tian S, Tang R, Marigowda G, Waltz D, Pilewski J; VX14-809-106 Investigator Group. Lumacaftor/ivacaftor in patients with cystic fibrosis and advanced lung disease homozygous for F508del-CFTR. J Cyst Fibros. 2018 Mar;17(2):228-235. doi: 10.1016/j.jcf.2017.09.012. Epub 2017 Nov 8. PMID 29126871

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 46 participants were enrolled and treated in the study.
Groups:
- LUM/IVA: Participants received lumacaftor (LUM) 400 milligram (mg) in combination with ivacaftor (IVA) 250 mg as fixed-dose combination (FDC) tablet orally every 12 hours (q12h) for 24 weeks. A reduced initial dose of LUM 200 mg in combination with IVA 125 mg FDC tablet orally q12h was permitted.
Period: Overall Study
Arm/Group | LUM/IVA
Started | 46
Completed | 33
Not Completed | 13
Not completed — Death | 1
Not completed — Physician Decision | 1
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Groups:
- LUM/IVA: Participants received LUM 400 mg in combination with IVA 250 mg as FDC tablet orally q12h for 24 weeks. A reduced initial dose of LUM 200 mg in combination with IVA 125 mg FDC tablet orally q12h was permitted.
Arm/Group | LUM/IVA
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: AE: any untoward medical occurrence in a participant during the study; event does not necessarily have a causal relationship with treatment. This includes any newly occurring event/previous condition that has increased in severity/frequency after informed consent form is signed. AE includes serious as well as non-serious AEs. SAE (subset of AE): medical event, which falls into any of the following categories, regardless of its relationship to study drug: death, life threatening adverse experience, in-patient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. TEAEs: AEs that started/ worsened on/after the start of study drug through the Safety Follow up Visit (4 weeks after the last dose of study drug). Results were reported as planned, as a combined single LUM/IVA arm irrespective of permitted dose modification.
Time Frame: Day 1 up to Week 28
Population: Safety Set included all participants who were exposed to any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LUM/IVA
Number analyzed (Participants) | 46
Participants
  Participants with AEs | 43
  Participants with SAEs | 18

2. Secondary Outcome: Absolute Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) Up to Week 24
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Hankinson and Wang standards were used to calculate percent predicted FEV1 (for age, gender, and height). The Hankinson standard was used for male participants 18 years and older and female participants 16 years and older. The Wang standard was used for male participants aged 12 to 17 years and for female participants aged 12 to 15 years. Results were reported as planned, as a combined single LUM/IVA arm irrespective of permitted dose modification.
Time Frame: Baseline, Up to Week 24
Population: Full Analysis Set (FAS) included all participants who were enrolled and administered any amount of study drug. Here, "Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent predicted of FEV1
Arm/Group | LUM/IVA
Number analyzed (Participants) | 32
Percent predicted of FEV1 | -0.4 (0.7)

3. Secondary Outcome: Absolute Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) Up to Week 24
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Hankinson and Wang standards were used to calculate FEV1 (for age, gender, race, and height). The Hankinson standard was used for male participants 18 years and older and female participants 16 years and older. The Wang standard was used for male participants aged 12 to 17 years and for female participants aged 12 to 15 years. Results were reported as planned, as a combined single LUM/IVA arm irrespective of permitted dose modification.
Time Frame: Baseline, Up to Week 24
Population: FAS included all participants who were enrolled and administered any amount of study drug. Here, "Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Liter (L)
Arm/Group | LUM/IVA
Number analyzed (Participants) | 32
Liter (L) | -0.02 (0.03)

4. Secondary Outcome: Duration For Which Participants Received Intravenous (IV) Antibiotics
Description: The duration for which participants received IV antibiotics for sinopulmonary signs and symptoms were reported. Results were reported as planned, as a combined single LUM/IVA arm irrespective of permitted dose modification.
Time Frame: Baseline through Week 24
Population: FAS included all participants who were enrolled and administered any amount of study drug. Here, "Number of Participants Analyzed" signifies those participants who received at least one IV antibiotic for sinopulmonary signs and symptoms.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | LUM/IVA
Number analyzed (Participants) | 22
Days | 11.38 (18.15)

5. Secondary Outcome: Number of Hospitalizations
Description: Number of hospitalizations (all causes) through Week 24 was summarized. Results were reported as planned, as a combined single LUM/IVA arm irrespective of permitted dose modification.
Time Frame: Baseline through Week 24
Population: as for outcome 3
Measure: Number; unit: Hospitalizations
Arm/Group | LUM/IVA
Number analyzed (Participants) | 16
Hospitalizations | 23

6. Secondary Outcome: Absolute Change From Baseline in Sweat Chloride at Average of Day 15 and Week 4
Description: Sweat samples were collected using an approved collection device. Baseline was defined as the average of the measurements at screening and on Day 1 pre-dose. The average absolute change from baseline in sweat chloride was derived as: (Average of Day 15 and Week 4 value) minus Baseline value. Results were reported as planned, as a combined single LUM/IVA arm irrespective of permitted dose modification.
Time Frame: Baseline, Day 15 and Week 4
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Millimoles per litre (mmol/L)
Arm/Group | LUM/IVA
Number analyzed (Participants) | 41
Millimoles per litre (mmol/L) | -16.4 (1.3)

7. Secondary Outcome: Absolute Change From Baseline in Cystic Fibrosis Questionnaire - Revised (CFQ-R) Respiratory Domain Score Through Week 24
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms (for example, coughing, congestion, wheezing), the scaled score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life. Results were reported as planned, as a combined single LUM/IVA arm irrespective of permitted dose modification.
Time Frame: Baseline, Through Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | LUM/IVA
Number analyzed (Participants) | 44
Units on a scale | 2.5 (1.7)

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 28
Description: AEs were reported as planned, as a combined single LUM/IVA arm irrespective of permitted dose modification.
Arm/Group | LUM/IVA
All-Cause Mortality (participants affected / at risk) | 1/46
Serious Adverse Events (participants affected / at risk) | 18/46
Other Adverse Events (participants affected / at risk) | 43/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LUM/IVA (N=46)
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1
Neuralgia (Nervous system disorders) | 1
Pyrexia (General disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 16
Bacteraemia (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LUM/IVA (N=46)
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Seasonal allergy (Immune system disorders) | 2
Drug hypersensitivity (Immune system disorders) | 1
Fatigue (General disorders) | 7
Chest pain (General disorders) | 4
Pain (General disorders) | 3
Pyrexia (General disorders) | 3
Asthenia (General disorders) | 1
Insomnia (Psychiatric disorders) | 4
Affect lability (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Irritability (Psychiatric disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Pulmonary function test decreased (Investigations) | 3
Blood glucose increased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 2
Blood creatine phosphokinase increased (Investigations) | 1
Blood glucose decreased (Investigations) | 1
Blood immunoglobulin E increased (Investigations) | 1
Blood phosphorus decreased (Investigations) | 1
Blood pressure diastolic increased (Investigations) | 1
Forced expiratory volume decreased (Investigations) | 1
Fungal test positive (Investigations) | 1
Oxygen consumption increased (Investigations) | 1
Prostatic specific antigen increased (Investigations) | 1
Sputum abnormal (Investigations) | 1
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Palpitations (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Headache (Nervous system disorders) | 7
Lethargy (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 1
Lacrimation increased (Eye disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal tract mucosal discolouration (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Nephrocalcinosis (Renal and urinary disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 20
Nasopharyngitis (Infections and infestations) | 3
Gastroenteritis viral (Infections and infestations) | 2
Vulvovaginal mycotic infection (Infections and infestations) | 2
Chronic sinusitis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Labyrinthitis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Sinusitis bacterial (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction Description: PI is free to publish results of the study after (1)first multi-center publication, (2)if sponsor elects not to publish the results, or (3)18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days(which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.